CLINICAL TRIAL: NCT04024033
Title: Effects of Pine Cone Extract on Serum IgE Levels in Perennial Rhinitis
Acronym: PCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of South Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pine Cone Extract
Record Dates: First submitted 2012-06-07; First posted 2019-07-18 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2022-11

CONDITIONS: Perennial Allergic Rhinitis
Keywords: perennial allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — PC6 extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- capsule (Active Comparator): patinets receiveing pine cone extract tablets
  Interventions: Dietary Supplement: pine cone extract
- placebo capsule (Placebo Comparator): patinets receiving placebo
  Interventions: Other: placebo

INTERVENTIONS:
Dietary Supplement: pine cone extract — pine cone extract capsule
  Arms: capsule
Other: placebo — placebo capsule
  Arms: placebo capsule

SUMMARY:
The medicinal properties of pinecones have been used for years to treat a variety of illnesses. In the mouse model, an extract of pine cones, poly-phenylpropanoid-polysaccharide complex (PPC), has been shown to reduce total serum IgE levels as well as decreased production of IL-4, a cytokine associated with allergic disease. In this study, the investigators aim to determine the effects that PPC will have on total serum IgE levels in adult subjects with perennial rhinitis.

DETAILED DESCRIPTION:
The study will be a parallel two-arm, double-blind design. The 80% power calculation was based upon preliminary data showing a greater than 30% reduction of total serum IgE in PPC recipients. This power calculation concluded that each arm will need a population of 18 subjects. These subjects will be recruited from a clinical practice of 4 academic allergists/immunologists. Seasonal allergy information will be recorded but the data will be analyzed for each group without any correction for seasonal effects.

Recruited subjects will sign the consent form, undergo a complete physical exam, and have skin testing repeated if historical skin tests data within three years is unavailable. The historical skin tests must have been performed using the same techniques as those used in the study. A prick skin test method using commercially available extracts will be used and the results graded according to standard criteria with measurements of the wheal and flare compared to the results of a positive control with histamine and a negative control of saline. A positive skin test will be defined as a wheal diameter 3 mm larger than the negative control with a flare of greater than or equal to 10 mm.

A nasal mucosal sample will also be obtained from the inferior turbinate with a plastic device (rhinoprobe). This sample will be frozen at the time of collection for future analysis. This procedure will be optional for subjects; if they consent it will be performed at each visit After screening, patients will be randomized to either of the two arms (placebo, or 32mg PPC/d). Patients will be instructed to take one capsule via oral route daily for 8 weeks. Subjects will be treated for two months with measurements of total serum IgE at the initial screening/randomization visit and following two months of treatment. Physical examination will be repeated at each visit. A variance of 5 days will be permitted for follow-up visits.

Rescue treatment with oral, non-sedating antihistamine will be permitted and number of doses will be recorded at each follow up visit. No nasal sprays will be allowed during the study. If symptoms are extreme, the study subject will be discontinued from the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with perennial allergic rhinitis with or without seasonal allergic rhinitis
2. Male or female participants must be 18 years of age or older

Exclusion Criteria:

1. Subjects receiving subcutaneous allergen immunotherapy or monoclonal anti-IgE (omalizumab)
2. Subject with hypersensitivity to PPC
3. Pregnant subjects (lactating post-partum women will be allowed to participate)
4. Subjects who are unable to cooperate/comply with study procedures or communicate with investigator in order to successfully complete the study
5. Subjects with severe skin disorders such as atopic dermatitis, dermatographism, psoriasis who could not have allergy skin testing and who have no prior skin testing completed within 3 years
6. Subjects with an infirmity, disability, or geographical location which seems likely to prevent regular attendance for patient visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-03 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Primary Objective ( total serum IgE) | 8 weeks
  To provide the proof-of-concept that daily administration of Immune Extra ™(each capsule with 16 mg total pine cone extract or 6 mg of PPC) reduces total serum IgE in subjects with rhinitis and sensitivity to perennial allergens, including dust mite (Dermatophagoides pteronyssinus and Dermatophagoides farinae), cockroach, cat, and dog.

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Ledford, M.D., Principal Investigator — Division of Allergy and Immunology, USF
Locations (1):
- Usf Asthma Allergy and Immunology Cru, Tampa, Florida, United States